CLINICAL TRIAL: NCT07210840
Title: Comparison Between Traditional Vestibular Rehabilitation Therapy And Virtual Reality In Management Of Patients With Chronic Dizziness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noran Kamal Gaber Hamdan, residant doctor at Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TVRT vs Virtual Reality Dizzin
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Chronic Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Traditional Vestibular Rehabilitation Therapy
  Interventions: Procedure: Traditional Vestibular Rehabilitation Therapy
- Group B (Active Comparator): Virtual Reality treatment
  Interventions: Procedure: Virtual Reality treatment

INTERVENTIONS:
Procedure: Virtual Reality treatment — Exercises delivered via a VR system simulating balance tasks and environments
  Arms: Group B
Procedure: Traditional Vestibular Rehabilitation Therapy — Customized vestibular exercises (gaze stabilization, balance, habituation, gait training).
  Arms: Group A

SUMMARY:
Chronic dizziness is a common and often debilitating condition, especially among older adults. It typically presents as a persistent sensation of unsteadiness, spinning, or motion lasting weeks or months. Most cases stem from vestibular system disorders, such as vestibular neuritis, benign paroxysmal positional vertigo (BPPV), Menière's disease, and bilateral vestibulopathy [1,2]. Symptoms may persist beyond the acute phase due to the brain's incomplete adaptation or maladaptive behaviors, like avoiding movement. Psychological factors, such as anxiety and stress, can worsen or prolong symptoms [3].

While many vestibular disorders resolve over time, some patients experience chronic symptoms due to poor central compensation or fear-based movement avoidance [2]. Chronic dizziness significantly impacts daily life-leading to imbalance, increased fall risk, reduced mobility, and emotional distress. Proper management is crucial to improving safety, independence, and quality of life [4].

Initial treatments may include medications or maneuvers like the Epley technique for BPPV. If symptoms persist, Vestibular Rehabilitation Therapy (VRT) is often recommended. VRT is a personalized exercise program aimed at enhancing the brain's ability to adapt, habituate, or compensate through substitution [6-8].

Recently, Virtual Reality (VR) has emerged as an innovative tool in vestibular rehab. It provides engaging, interactive environments for practicing balance and visual-vestibular tasks. Studies suggest that VR is feasible, well-tolerated, and effective, particularly for patients with persistent or visually-induced dizziness [9,10].

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged 18-70 years.

  * Patients diagnosed with chronic dizziness (duration >3 months) due to peripheral vestibular disorders (e.g., vestibular neuritis, BPPV, unilateral vestibular hypofunction).

Exclusion Criteria:

* Presence of central vestibular disorders (e.g., multiple sclerosis, cerebellar ataxia,

  * stroke).
  * Patients in acute phase
  * Presence of severe visual impairment
  * Presence of motor disabilities that prevent safe participation in rehabilitation exercises.
  * Cognitive impairment or psychiatric illness that decrease ability to follow instructions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
cure rate | baseline
  the clinical effectiveness of treatment in management of patients with chronic dizziness due to vestibular disorders.